CLINICAL TRIAL: NCT06545513
Title: The Prevalence of Depression and Anxiety Among Chronic Pain Patients in the Netherlands
Brief Title: Depression and Anxiety Among Chronic Pain Patients in the Netherlands
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Marlies Smits, MD, Amsterdam UMC, location VUmc
Other Study IDs: 2022.0372
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Depression, Anxiety
Keywords: Chronic pain; Depression; Anxiety
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with chronic pain: The patients have completed surveys prior or during their visit at the chronic pain outpatient clinic.

SUMMARY:
The aim of this study is to examine the prevalence of anxiety and depression among patients with chronic pain attending secondary and tertiary pain clinics in the Netherlands. Additionally, the study explores how pain intensity, sociodemographic factors, and the presence of anxiety or depression are associated with quality of life in this population.

Using an anonymized dataset provided by the data manager, we aimed to prevent a low response rate at Amsterdam UMC and thereby reduce the risk of non-response bias.

DETAILED DESCRIPTION:
Chronic pain is defined as pain which exists for a period longer than 3 months. The prevalence of chronic pain in the Netherlands is estimated to be 19 percent. Chronic pain is a complex disorder which is often challenging to treat. The dynamic interaction between de different aspects of chronic pain, like the somatic, physical and social aspects, make the treatment challenging. Patients with chronic pain have a three times increased risk of developing psychiatric symptoms (usually mood and anxiety disorders) and vice versa, patients with depression have a three times increased risk of developing chronic pain. Also independently chronic pain and depression are both invalidating disorders, regardless of age and gender. It has been found that there is an increased risk of suicide among patients with chronic pain. The complex interaction between chronic pain and depression and their cumulative effect on the quality of life in the Netherlands has not yet been completely identified. This is because the interaction between chronic pain and depression is not yet fully understood. The treatment can be improved when the interaction between pain and depression is better understood.

The research acts as a preliminary investigation for the treatment of patients with chronic pain with intrvenous esketamine, a recently approved treatment for treatment resistant depression.

ELIGIBILITY:
Patients over 18 years old with chronic pain, who have been treated at the pain clinic at Amsterdam UMC from 2020 to 2024, will be included in the study, provided they have completed the HADS questionnaires in full. Patients with incomplete HADS questionnaires and those who have filed a general objection to the use of their data for this scientific research will be excluded from participation in the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain under treatment at chronic pain outpatient clinics at Amsterdam UMC.
Sampling Method: Non-Probability Sample
Enrollment: 3240 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression | 2020-2024
  prevalence of depression among chronic pain patients

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Magni G, Marchetti M, Moreschi C, Merskey H, Luchini SR. Chronic musculoskeletal pain and depressive symptoms in the National Health and Nutrition Examination. I. Epidemiologic follow-up study. Pain. 1993 May;53(2):163-168. doi: 10.1016/0304-3959(93)90076-2. PMID 8336986
- [Background] Carroll LJ, Cassidy JD, Cote P. Depression as a risk factor for onset of an episode of troublesome neck and low back pain. Pain. 2004 Jan;107(1-2):134-9. doi: 10.1016/j.pain.2003.10.009. PMID 14715399
- [Background] Racine M. Chronic pain and suicide risk: A comprehensive review. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Dec 20;87(Pt B):269-280. doi: 10.1016/j.pnpbp.2017.08.020. Epub 2017 Aug 26. PMID 28847525
- See also: International Classification of Disease (11th version) — https://icd.who.int/browse/2024-01/mms/en